CLINICAL TRIAL: NCT03395756
Title: Investigation of the Potential for Intramuscular Depot Medroxyprogesterone Acetate as Emergency Contraception
Brief Title: Depot Medroxyprogesterone Acetate as Emergency Contraception
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Brian T. Nguyen, MD MSc, Assistant Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS-17-01006
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Emergency Contraception; Contraception
Keywords: Depot Medroxyprogesterone acetate; Injectable birth control
MeSH Terms: interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Intervention Model Description: Participants in this study will be assigned to one of three groups based on leading follicle size: 12-14 mm, 15-17mm, and 18 mm or greater. Each group will receive the same medication (intramuscular depot medroxyprogesterone acetate), and be followed in the same manner for five consecutive days after administration with transvaginal ultrasound and blood draws for hormonal assays (progesterone, estradiol, and luteinizing hormone levels)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 12-14 mm follicle size group (Active Comparator): Once the participant's leading follicle reaches 12-14mm, she will receive an IM administration of 150 mg Depot-Medroxyprogesterone Acetate. Prior to administration, she will have blood drawn for baseline progesterone, estradiol, and LH levels. One hour after receiving the injection, she will have blood drawn for medroxyprogesterone acetate levels. The next day, she will undergo a transvaginal ultrasound to assess the leading follicle and will have blood drawn for progesterone, estradiol, LH, and medroxyprogesterone acetate levels. For the next 4 consecutive days, she will have daily transvaginal ultrasounds to assess for signs of follicular rupture, and blood draws for hormonal assays. After, she will return twice weekly for two weeks for blood draw for progesterone levels.
  Interventions: Drug: Depot-Medroxyprogestereone Acetate
- 15-17 mm follicle size group (Active Comparator): Once the participant's leading follicle reaches 15-17mm, she will receive an IM administration of 150 mg Depot-Medroxyprogesterone Acetate. Prior to administration, she will have blood drawn for baseline progesterone, estradiol, and LH levels. One hour after receiving the injection, she will have blood drawn for medroxyprogesterone acetate levels. The next day, she will undergo a transvaginal ultrasound to assess the leading follicle and will have blood drawn for progesterone, estradiol, LH, and medroxyprogesterone acetate levels. For the next 4 consecutive days, she will have daily transvaginal ultrasounds to assess for signs of follicular rupture, and blood draws for hormonal assays. After, she will return twice weekly for two weeks for blood draw for progesterone levels.
  Interventions: Drug: Depot-Medroxyprogestereone Acetate
- 18 mm or greater follicle size group (Active Comparator): Once the participant's leading follicle reaches 18mm or greater, she will receive an IM administration of 150 mg Depot-Medroxyprogesterone Acetate. Prior to administration, she will have blood drawn for baseline progesterone, estradiol, and LH levels. One hour after receiving the injection, she will have blood drawn for medroxyprogesterone acetate levels. The next day, she will undergo a transvaginal ultrasound to assess the leading follicle and will have blood drawn for progesterone, estradiol, LH, and medroxyprogesterone acetate levels. For the next 4 consecutive days, she will have daily transvaginal ultrasounds to assess for signs of follicular rupture, and blood draws for hormonal assays. After, she will return twice weekly for two weeks for blood draw for progesterone levels.
  Interventions: Drug: Depot-Medroxyprogestereone Acetate

INTERVENTIONS:
Drug: Depot-Medroxyprogestereone Acetate — Administration of 150 mg intramuscular depot medroxyprogesterone acetate

SUMMARY:
Background:

The prevalence of repeat unprotected intercourse after EC use in the same cycle demonstrate the need for more self-bridging emergency contraceptive options. We propose the use of intramuscular Depot Medroxyprogesterone acetate (DMPA) as EC, which has been shown to inhibit follicular activity within 24 hours, and provide on-going contraception via suppression or disruption of ovulation.

Objective:

The objective of this study is to explore the potential of depot medroxyprogesterone acetate (DMPA) given as a 150-mg intramuscular injection for use as an emergency contraceptive.

Study population:

Healthy regularly menstruating women aged 18-39 years old will be invited to participate if they fulfill inclusion criteria. The participants will undergo a screening visit during the midluteal phase of their cycle, and will be enrolled if a serum progesterone level is >3ng/ml.

Methodology:

Participants will be assigned to one of three groups based on leading follicle size. Starting cycle Day 8, transvaginal ultrasounds will be performed to assess the size of the leading follicle. Once the follicle has reached the pre-assigned size, 150 mg IM DMPA will be administered. Blood will be collected for baseline hormonal assays. For 5 consecutive days, daily blood will be drawn for hormonal assays and daily transvaginal ultrasound will be performed to assess for signs of ovulation. The participant will then return for twice weekly progesterone levels for 2 weeks for study completion.

DETAILED DESCRIPTION:
The proposed study will enroll 36 healthy, non-pregnant, non-breastfeeding, reproductive age women with regular ovulatory cycles. Potential participants will undergo screening, which will include a history, physical exam, assessment of vital signs, and blood draw for assessment of ovulation via mid-luteal progesterone levels. If her progesterone level confirms ovulatory status (> 3 ng/ml), she will be offered enrollment and assigned to one of three follicular phase groups based on her leading follicle size in the next cycle: 12-14 mm, 15-17 mm, and ≥18 mm. To determine follicle size, participants will receive serial transvaginal ultrasound (TVUS) scans of their ovarian follicles starting on cycle day 8 of the next menstrual cycle. The scans will be performed three times weekly to identify her leading follicle. Once the leading follicle has reached its assigned size, DMPA will be administered. Blood samples will be obtained prior to administration for baseline hormonal assays. One hour after administration, blood will be drawn for MPA levels. For the following five consecutive days, the participant will undergo daily TVUS to detect signs of follicular rupture and blood draws to assess serum markers of ovulation (estradiol, progesterone, and luteinizing hormone). On the first day, 24 hours after DMPA administration, blood will be drawn for MPA levels as well. After five days, the participant will return twice weekly for two weeks to provide serum progesterone levels to detect any delayed ovulation or ovulatory dysfunction. At the final visit, she will fill out a simple survey to assess her satisfaction with DMPA as an EC method, and whether she would recommend this method to others.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of reproductive age (18-39 years old) with BMI 18-30 kg/m2
* Regular menses for the last 3 months
* Cycle duration 24 to 35 days
* Women using copper IUD, sterilization, or barrier methods as current or preferred birth control method, and women reporting exclusive sex with women
* English- or Spanish-speaking

Exclusion Criteria:

* Any contraindications to progesterone contraception per teh CDC Medical Eligibility Criteria (Category 3 or 4)
* On medications that can alter, or be altered by, progesterone contraceptive steroid hormone (e.g., aminoglutethimide or other anti-steroid medication)
* Use of any hormonal contraceptive pill, patch, or vaginal ring in the month prior to recruitment
* Use of depot-medroxyprogesterone acetate in teh 10 months prior to recruitment
* Currently pregnant and/or breastfeeding
* History of allergic reaction to depot medroxyprogesterone acetate (rash, urticaria, anaphylaxis)

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Ovulation | 5 days to 3 weeks
  Follicle rupture on ultrasound preceded by LH surge 21 IU/L or greater, followed by progesterone level 3 ng/ml or greater.
Ovulation Suppression | 5 days to 3 weeks
  Lack of follicular rupture on ultrasound with or without appropriate LH surge of 21 IU/L or greater and without elevation in progesterone levels to 3 ng/ml or greater
Ovulatory dysfunction | 5 days to 3 weeks
  Rupture of leading follicle without appropriate LH surge (less than 21 IU/L) and without appropriate progesterone elevation after rupture (less then 3 ng/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn L Schickler, MD, Principal Investigator — University of Southern California; Brian Nguyen, MD, MSCP, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California Keck Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daniels K, Jones J, Abma J. Use of emergency contraception among women aged 15-44: United States, 2006-2010. NCHS Data Brief. 2013 Feb;(112):1-8. PMID 23742711
- [Background] ESHRE CapriWorkshop Group. Emergency contraception. Widely available and effective but disappointing as a public health intervention: a review. Hum Reprod. 2015 Apr;30(4):751-60. doi: 10.1093/humrep/dev019. Epub 2015 Feb 11. PMID 25678571
- [Background] Glasier A, Cameron ST, Blithe D, Scherrer B, Mathe H, Levy D, Gainer E, Ulmann A. Can we identify women at risk of pregnancy despite using emergency contraception? Data from randomized trials of ulipristal acetate and levonorgestrel. Contraception. 2011 Oct;84(4):363-7. doi: 10.1016/j.contraception.2011.02.009. Epub 2011 Apr 2. PMID 21920190
- [Background] Turok DK, Gurtcheff SE, Handley E, Simonsen SE, Sok C, North R, Frost C, Murphy PA. A survey of women obtaining emergency contraception: are they interested in using the copper IUD? Contraception. 2011 May;83(5):441-6. doi: 10.1016/j.contraception.2010.08.011. Epub 2010 Sep 29. PMID 21477687
- [Background] Mishell DR Jr. Pharmacokinetics of depot medroxyprogesterone acetate contraception. J Reprod Med. 1996 May;41(5 Suppl):381-90. PMID 8725700
- [Background] Ortiz A, Hirol M, Stanczyk FZ, Goebelsmann U, Mishell DR. Serum medroxyprogesterone acetate (MPA) concentrations and ovarian function following intramuscular injection of depo-MPA. J Clin Endocrinol Metab. 1977 Jan;44(1):32-8. doi: 10.1210/jcem-44-1-32. PMID 833262
- [Background] Fotherby K, Koetsawang S, Mathrubutham M. Pharmacokinetic study of different doses of Depo Provera. Contraception. 1980 Nov;22(5):527-36. doi: 10.1016/0010-7824(80)90105-5. PMID 6451351
- [Background] Petta CA, Faundes A, Dunson TR, Ramos M, DeLucio M, Faundes D, Bahamondes L. Timing of onset of contraceptive effectiveness in Depo-Provera users. II. Effects on ovarian function. Fertil Steril. 1998 Nov;70(5):817-20. doi: 10.1016/s0015-0282(98)00309-4. PMID 9806559
- [Background] Croxatto HB, Brache V, Pavez M, Cochon L, Forcelledo ML, Alvarez F, Massai R, Faundes A, Salvatierra AM. Pituitary-ovarian function following the standard levonorgestrel emergency contraceptive dose or a single 0.75-mg dose given on the days preceding ovulation. Contraception. 2004 Dec;70(6):442-50. doi: 10.1016/j.contraception.2004.05.007. PMID 15541405
- [Background] Shen J, Che Y, Showell E, Chen K, Cheng L. Interventions for emergency contraception. Cochrane Database Syst Rev. 2017 Aug 2;8(8):CD001324. doi: 10.1002/14651858.CD001324.pub5. PMID 28766313
- [Background] Wilcox AJ, Weinberg CR, Baird DD. Timing of sexual intercourse in relation to ovulation. Effects on the probability of conception, survival of the pregnancy, and sex of the baby. N Engl J Med. 1995 Dec 7;333(23):1517-21. doi: 10.1056/NEJM199512073332301. PMID 7477165
- [Background] Long-term reversible contraception. Twelve years of experience with the TCu380A and TCu220C. Contraception. 1997 Dec;56(6):341-52. PMID 9494767
- [Background] Harper CC, Speidel JJ, Drey EA, Trussell J, Blum M, Darney PD. Copper intrauterine device for emergency contraception: clinical practice among contraceptive providers. Obstet Gynecol. 2012 Feb;119(2 Pt 1):220-6. doi: 10.1097/AOG.0b013e3182429e0d. PMID 22270272
- [Background] Wu S, Godfrey EM, Wojdyla D, Dong J, Cong J, Wang C, von Hertzen H. Copper T380A intrauterine device for emergency contraception: a prospective, multicentre, cohort clinical trial. BJOG. 2010 Sep;117(10):1205-10. doi: 10.1111/j.1471-0528.2010.02652.x. Epub 2010 Jul 7. PMID 20618314
- [Background] Rowe P, Farley T, Peregoudov A, Piaggio G, Boccard S, Landoulsi S, Meirik O; IUD Research Group of the UNDP/UNFPA/WHO/World Bank Special Programme of Research; Development and Research Training in Human Reproduction. Safety and efficacy in parous women of a 52-mg levonorgestrel-medicated intrauterine device: a 7-year randomized comparative study with the TCu380A. Contraception. 2016 Jun;93(6):498-506. doi: 10.1016/j.contraception.2016.02.024. Epub 2016 Feb 23. PMID 26916172
- [Background] Royer PA, Turok DK, Sanders JN, Saltzman HM. Choice of Emergency Contraceptive and Decision Making Regarding Subsequent Unintended Pregnancy. J Womens Health (Larchmt). 2016 Oct;25(10):1038-1043. doi: 10.1089/jwh.2015.5625. Epub 2016 Mar 31. PMID 27032057
- [Background] Novikova N, Weisberg E, Stanczyk FZ, Croxatto HB, Fraser IS. Effectiveness of levonorgestrel emergency contraception given before or after ovulation--a pilot study. Contraception. 2007 Feb;75(2):112-8. doi: 10.1016/j.contraception.2006.08.015. Epub 2006 Oct 27. PMID 17241840
- [Background] Jones J, Mosher W, Daniels K. Current contraceptive use in the United States, 2006-2010, and changes in patterns of use since 1995. Natl Health Stat Report. 2012 Oct 18;(60):1-25. PMID 24988814
- [Background] Trussell J. Contraceptive failure in the United States. Contraception. 2011 May;83(5):397-404. doi: 10.1016/j.contraception.2011.01.021. Epub 2011 Mar 12. PMID 21477680
- [Background] Sundaram A, Vaughan B, Kost K, Bankole A, Finer L, Singh S, Trussell J. Contraceptive Failure in the United States: Estimates from the 2006-2010 National Survey of Family Growth. Perspect Sex Reprod Health. 2017 Mar;49(1):7-16. doi: 10.1363/psrh.12017. Epub 2017 Feb 28. PMID 28245088
- [Background] Curtis KM, Tepper NK, Jatlaoui TC, Berry-Bibee E, Horton LG, Zapata LB, Simmons KB, Pagano HP, Jamieson DJ, Whiteman MK. U.S. Medical Eligibility Criteria for Contraceptive Use, 2016. MMWR Recomm Rep. 2016 Jul 29;65(3):1-103. doi: 10.15585/mmwr.rr6503a1. PMID 27467196
- [Background] Gemzell-Danielsson K, Berger C, P G L L. Emergency contraception -- mechanisms of action. Contraception. 2013 Mar;87(3):300-8. doi: 10.1016/j.contraception.2012.08.021. Epub 2012 Oct 29. PMID 23114735
- [Background] Siriwongse T, Snidvongs W, Tantayaporn P, Leepipatpaiboon S. Effect of depo-medroxyprogesterone acetate on serum progesterone levels when administered on various cycle days. Contraception. 1982 Nov;26(5):487-93. doi: 10.1016/0010-7824(82)90147-0. PMID 6218964
- [Background] Curtis KM, Jatlaoui TC, Tepper NK, Zapata LB, Horton LG, Jamieson DJ, Whiteman MK. U.S. Selected Practice Recommendations for Contraceptive Use, 2016. MMWR Recomm Rep. 2016 Jul 29;65(4):1-66. doi: 10.15585/mmwr.rr6504a1. PMID 27467319
- [Background] Croxatto HB, Fuentealba B, Brache V, Salvatierra AM, Alvarez F, Massai R, Cochon L, Faundes A. Effects of the Yuzpe regimen, given during the follicular phase, on ovarian function. Contraception. 2002 Feb;65(2):121-8. doi: 10.1016/s0010-7824(01)00299-2. PMID 11927114
- [Background] Croxatto HB, Brache V, Massai R, Alvarez F, Forcelledo ML, Pavez M, Cochon L, Salvatierra AM, Faundes A. Feasibility study of Nestorone-ethinylestradiol vaginal contraceptive ring for emergency contraception. Contraception. 2006 Jan;73(1):46-52. doi: 10.1016/j.contraception.2005.06.071. Epub 2005 Nov 14. PMID 16371294
- [Background] Duijkers IJ, Louwe LA, Braat DD, Klipping C. One, two or three: how many directions are useful in transvaginal ultrasound measurement of ovarian follicles? Eur J Obstet Gynecol Reprod Biol. 2004 Nov 10;117(1):60-3. doi: 10.1016/j.ejogrb.2004.01.005. PMID 15474246
- [Background] Pardthaisong T, Gray RH. In utero exposure to steroid contraceptives and outcome of pregnancy. Am J Epidemiol. 1991 Oct 15;134(8):795-803. doi: 10.1093/oxfordjournals.aje.a116152. PMID 1835282
- [Background] Pardthaisong T, Gray RH, McDaniel EB, Chandacham A. Steroid contraceptive use and pregnancy outcome. Teratology. 1988 Jul;38(1):51-8. doi: 10.1002/tera.1420380108. PMID 2845595
- [Background] Pardthaisong T, Yenchit C, Gray R. The long-term growth and development of children exposed to Depo-Provera during pregnancy or lactation. Contraception. 1992 Apr;45(4):313-24. doi: 10.1016/0010-7824(92)90053-v. PMID 1387602